CLINICAL TRIAL: NCT00795262
Title: A 22-week Randomized, Cross-over Study Comparing the Effects of Quinapril and Quinapril Plus Alpha-lipoic Acid (ALA) on Patients With Diabetes Mellitus and Hypertension
Brief Title: Effects of Quinapril 40 mg With Alpha Lipoic Acid or Placebo on Diabetes and Hypertension
Acronym: QUALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InVasc Therapeutics, Inc. (Industry)
Responsible Party: Syed T. Rahman, MD, Atlanta Vascular Research Foundation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV-064 QUALITY
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes; Hypertension
Keywords: brachial artery reactivity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Quinapril; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo comparator (Placebo Comparator): Quinapril 40 mg (Accupril)plus placebo will be given for 8 weeks.
  Interventions: Drug: accupril, placebo
- Active comparator (Active Comparator): Quinapril 40 mg plus Alpha Lipoic Acid (ALA)on vascular effects of patients with diabetes and hypertension
  Interventions: Drug: Quinapril (Accupril) plus Alpha Lipoic Acid; Drug: accupril, alpha lipoic acid

INTERVENTIONS:
Drug: Quinapril (Accupril) plus Alpha Lipoic Acid — Patients in Arm 2 (n=20) will receive quinapril 40 mg and Alpha Lipoic Acid (600 mg/day)for an 8-week treatment period (Treatment A).
  Other Names: ALA; Alpha Lipoic Acid; Quinapril; Accupril
  Arms: Active comparator
Drug: accupril, placebo — accupril 40 mg
  Other Names: Accupril; quinapril
  Arms: placebo comparator
Drug: accupril, alpha lipoic acid — accupril (quinapril) 40 mg plus alpha lipoic acid 600 mg
  Other Names: quinapril; accupril; ALA; alpha lipoic acid; lipoic acid
  Arms: Active comparator

SUMMARY:
We will evaluate the combination of quinapril and alpha lipoic acid in patients with diabetes mellitus and hypertension. We will determine whether the combination of quinapril and lipoic acid as compared to quinapril and placebo provides benefit on systemic blood pressure and proteinuria.

DETAILED DESCRIPTION:
The participant will be randomized to either quinapril 40 mg and alpha lipoic acid versus quinapril 40 mg and placebo for 8 weeks. There will be a wash out period of 4 weeks between the cross over. The participant will be assigned the cross over for 8 weeks on the opposite therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who have a diagnosis of diabetes mellitus as defined by fasting blood glucose levels greater than ot equal to 126mg/dL and a systolic BP greater than 125 mm Hg at the time of screening will be included in the study. Patients may be on antihypertensive medication but not on ACE inhibitor or ARB therapy at the time of enrollment.

Exclusion Criteria:

Systolic blood pressure > 180 mmHg Creatinine > 2.5 mg/dl Glycosylated hemoglobin > 7.5% Congestive heart failure (NYHA Class II, III or IV) Coronary angiography planned prior to baseline sampling Chronic autoimmune disease Chronic inflammatory disease or known cancer in evolution life expectancy < 1 year Immunosuppressives or treatment with any other investigational drug within the last 30 days Pregnant or nursing women Participants who experience any side effects to quinapril and/or alpha lipoic acid

Women of childbearing potential Women of childbearing potential enrolled in the study should use one of the acceptable methods of birth control as listed below

1. Abstinence, meaning a total lack of any sexual activity.
2. Oral contraceptives (the "pill"),
3. Contraceptive injections,
4. Intrauterine device,
5. Double-barrier method (diaphragm or condom + spermicidal cream),
6. Contraceptive patch, or
7. Male partner sterilization.

Pregnancy Any pregnancy that occurs during study participation must be reported to the Principal Investigator and the study coordinator at the earliest. The pregnancy must be followed up to determine outcome and status of the mother and child. To ensure subject safety, any subject that becomes pregnant during the study will be discontinued from the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Comparison of relative change of systolic BP/diastolic BP and urinary albumin excretion from baseline in diabetic patients treated with quinapril plus lipoic acid versus quinapril and placebo. | The total study period is 22 weeks i.e. the initial prescreening visit followed 1 week later by the baseline study visit, 8 weeks of treatment (Treatment A or B), 4 weeks washout, 8 weeks of treatment (Treatment A or B).

SECONDARY OUTCOMES:
Comparison of patients treated with quinapril plus lipoic acid versus quinapril plus placebo in the following areas: a) Changes from baseline in high sensitivity C-reactive protein, adiponectin, and leptin | at baseline (week-1), weeks 8, 12 and 20.

CONTACTS AND LOCATIONS:
Overall Officials: Syed T. Rahman, MD, Principal Investigator — Atlanta Vascular Research Foundation
Locations (1):
- Atlanta Vascular Research Foundation, Tucker, Georgia, United States